CLINICAL TRIAL: NCT03760978
Title: Efficacy and Safety of Dexmedetomidine for Prolonged Sedation in Pediatric Intensive Care Units
Brief Title: Dexmedetomidine for Prolonged Sedation in PICUs
Acronym: PROSDEX
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, angela amigoni, Principal Investigator, Azienda Ospedaliera di Padova
Other Study IDs: 4466/AO/18; AOP1403
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Prolonged Sedation
Keywords: sedation; dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dex group: Critically ill patients <18 year-old receiving prolonged sedation with endovenous dexmedetomidine (dosage 0.2 mcg/Kg/hour to 1.8 mcg/Kg/hour) more than 24 hours
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: dexdor; precedex

SUMMARY:
Sedation management of the critically ill patients is still a challenge for the pediatric intensivists. Worldwide the most common sedation approach includes the concomitant use of opioids and benzodiazepines. The use of these drugs is associated with adverse events contributing with morbidity, such as decreased spontaneous ventilation, withdrawal syndrome and delirium onset. Moreover, benzodiazepine demonstrated a neurotoxic apoptotic effect that could potentially impact neurocognitive outcome.

Dexmedetomidine (DEX) is a selective alpha-2-adrenergic agonist with sedative, analgesic and anxiolytic effects. Its unique pharmacological profile allows reaching a conscious sedation state with minimal respiratory depression, promoting faster ventilation weaning and better collaboration with the medical staff. Moreover, DEX seems to present adjuvant properties towards withdrawal syndrome and delirium. Finally, some studies in animals suggested that Dexmedetomidine might have a role of neuro-protection, especially in a contest of cerebral ischemia.

Currently, the Food and Drug Administration (FDA) and the European Medicines Agency (EMA) approved DEX only for the adult population and for sedation lasting not more than 24 hours. The Italian Medicines Agency (AIFA), in January 2016, approve DEX in children for specific indications including difficult sedation in mechanically ventilated critically ill patients. Up to now, few data are still available regarding its efficacy and safety for prolonged sedation in Pediatric Intensive Care Units (PICUs) and no studies have reported the use of DEX after AIFA's approval so far.

Aims of the study are:

to evaluate the characteristics of DEX use for prolonged sedation ≥24 hours in critically ill children (indication, dosages, time of infusion, time of infusion weaning, association with other drugs); to evaluate its efficacy in terms of comfort and conventional drug sparing, using standardized and validate measures; further, to evaluate its efficacy in terms of reduction of incidence of withdrawal syndrome and delirium; to evaluate its safety profile collecting any adverse event potentially correlated with its administration; to define if efficacy and safety could differ among approved indications versus not-approved ones.

Design: Multicenter observational prospective study, involving tertiary-care PICUs.

Study period: From January 2016 up to reaching of the calculated sample size (N patients =163).

Population: All critically ill patients <18 years who received prolonged sedation including DEX for ≥24 hours. In case of multiple infusions, only data regarding the first infusion will be included. Exclusion criteria: extreme prematurity (<28 weeks of gestational age), hypersensitivity to the active substance, incomplete data form. .

Collecting data strategy: Data will be prospectively collected from each Institution by means of a anonymous standardized form completed by two different investigators per center. For each patient, the following variables will be collected:

demographics characteristics (age, gender, race, weight) and clinical features (main diagnosis, associated morbidities, PIM3 score ad admission, number of high intensity interventions during PICU-stay, mechanical ventilation features, inotropic drugs use, length of stay, survival at discharge); DEX administration characteristics (indication, loading dose, minimum and maximum dosages, duration of DEX infusion, duration of DEX infusion weaning) and information on concomitant use of analgesics or sedative drugs (name of drugs and respective dosages at DEX starting time and 24 hours later); clinical scores of analgesia and sedation (Comfort Behavior Scale, CBS), withdrawal syndrome (Withdrawal Assessment Toll-1, WAT-1) and delirium (Cornell Assessment of Pediatric Delirium, CAPD) depending on the respective indication, registered immediate pre-DEX and 24 hours later; any adverse event potentially related to DEX administration and any related intervention, if present. In particular, we the investigators evaluate if bradycardia, hypotension (with or without poor perfusion), hypertension, agitations or other events are registered during the infusion. Further, investigators will register if any sign of DEX withdrawal (tachycardia, hypertension, agitation, other) are present immediately after the infusion.

Statistical analysis: Descriptive and analytic statistics will be performed according with the variable characteristics. A causal multivariate model will be developed to identify any significant risk or protective factors towards adverse outcomes (ineffective sedation, onset of adverse events).

ELIGIBILITY:
Inclusion Criteria:

* age <18 years
* admission to PICU
* sedation with dexmedetomidine lasted more than 24 hours
* written informed consent

Exclusion Criteria:

* extreme prematurity (<28 weeks of gestational age)
* hypersensitivity to the active substance
* incomplete data regarding outcome measures

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Critically ill children admitted to PICU
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Comfort Behavior Scale (CBS) | Immediately before DEX start and 24 hours later
  Standardized validated score for sedation level and pain assessment; range 6-30; lower values represent a deep level of sedation

SECONDARY OUTCOMES:
Opioid and benzodiazepines dosage | Immediately before DEX start and 24 hours later.
  Opioid and benzodiazepines cumulative and maximal dosage

OTHER OUTCOMES:
Withdrawal Assessment Tool-1 | Immediately before DEX start and 24 hours later.
  Standardized validated score for the assessment of withdrawal syndrome; range 0-12; higher values represent a more severe withdrawal syndrome; withdrawal syndrome is probable if score is > 2
Cornell Assessment of Pediatric Delirium, CAPD | Immediately before DEX start and 24 hours later
  Standardized validated score for the assessment of pediatric delirium; range 0-32; higher scores represent a more severe presence of delirium; delirium is probable if score is > 8
Onset of adverse events | During and immediately after dexmedetomidine infusion.
  any adverse event potentially related with DEX-administration

CONTACTS AND LOCATIONS:
Overall Officials: angela amigoni, MD, Principal Investigator — Azienda Ospedaliera di Padova
Locations (9):
- Italy (9):
  - Pediatric Intensive Care Unit, Children's Hospital C.Arrigo, Alessandria, Italy, Alessandria
  - Pediatric Intensive Care Unit, ASST John XXIII Pope Hospital, Bergamo, Italy, Bergamo
  - Pediatric Intensive Care Unit, S.Orsola Malpighi Hospital, University of Bologna, Italy, Bologna
  - Pediatric Intensive Care Unit, Children's Hospital V.Buzzi, Milan, Italy, Milan
  - Pediatric and Neonatal Intensive Care Unit, Maggiore della Carità Hospital, Novara, Italy, Novara
  - Terapia Intensiva Pediatrica Azienda Ospedaliera di Padova, Padua
  - Pediatric Intensive Care Unit, Bambino Gesù Children's Hospital, Rome, Italy, Roma
  - Pediatric Intensive Care Unit, A.Gemelli Hospital, Sacro Cuore Catholic University, Rome Italy, Rome
  - Pediatric Intensive Care Unit, Burlo Garofalo Hospital, University of Trieste, Italy, Trieste

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mondardini MC, Astuto M, Amigoni A. Inclusion of dexmedetomidine for pediatric indications in the list of medicinal products issued by the National Law 648/96. Minerva Anestesiol. 2017 Aug;83(8):891-892. doi: 10.23736/S0375-9393.17.11975-9. Epub 2017 Mar 3. No abstract available. PMID 28256816
- [Result] Romagnoli S, Amigoni A, Blangetti I, Casella G, Chelazzi C, Forfori F, Garisto C, Mondardini MC, Moltrasio M, Pasero D, Principi T, Ricci Z, Tarantino F, Conti G. Light sedation with dexmedetomidine: a practical approach for the intensivist in different ICU patients. Minerva Anestesiol. 2018 Jun;84(6):731-746. doi: 10.23736/S0375-9393.18.12350-9. Epub 2018 Feb 5. PMID 29405671
- [Result] Sperotto F, Mondardini MC, Vitale F, Daverio M, Campagnano E, Ferrero F, Rossetti E, Vasile B, Dusio MP, Ferrario S, Savron F, Brugnaro L, Amigoni A; Pediatric Neurological Protection and Drugs (PeNPAD) Study Group. Prolonged sedation in critically ill children: is dexmedetomidine a safe option for younger age? An off-label experience. Minerva Anestesiol. 2019 Feb;85(2):164-172. doi: 10.23736/S0375-9393.18.13062-8. Epub 2018 Oct 30. PMID 30394067
- [Result] Grant MJ, Schneider JB, Asaro LA, Dodson BL, Hall BA, Simone SL, Cowl AS, Munkwitz MM, Wypij D, Curley MA; Randomized Evaluation of Sedation Titration for Respiratory Failure Study Investigators. Dexmedetomidine Use in Critically Ill Children With Acute Respiratory Failure. Pediatr Crit Care Med. 2016 Dec;17(12):1131-1141. doi: 10.1097/PCC.0000000000000941. PMID 27654816
- [Result] Tabacco B, Tacconi C, Amigoni A. Survey on monitoring analgesia and sedation in the Italian Pediatric Intensive Care Units. Minerva Anestesiol. 2017 Oct;83(10):1010-1016. doi: 10.23736/S0375-9393.17.11707-4. Epub 2017 Mar 28. PMID 28358177
- [Result] Mason KP, Lerman J. Review article: Dexmedetomidine in children: current knowledge and future applications. Anesth Analg. 2011 Nov;113(5):1129-42. doi: 10.1213/ANE.0b013e31822b8629. Epub 2011 Aug 4. PMID 21821507
- See also: see Group of Study PeNPAD (Italian Research Group on Pediatric Neurological Protection and Drugs) — http://www.sarnepi.it